CLINICAL TRIAL: NCT01232075
Title: Extended Letrozole Regimen Versus Clomiphene Citrate for Superovulation in Patients With Unexplained Infertility Undergoing Intrauterine Insemination
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Ahmed Elgazzar Hospital (Other)
Responsible Party: Usama Fouda,M.D, PhD, Cairo university
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: clomid/extended letr/unexp.inf
Record Dates: First submitted 2010-11-01; First posted 2010-11-02 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-07

CONDITIONS: Infertility
Keywords: Letrozole ,Clomiphene citrate , IUI,unexplained infertility
MeSH Terms: conditions — Infertility | interventions — Letrozole; Clomiphene

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Extended letrozole regimen (Experimental)
  Interventions: Drug: Extended letrozole regimen
- Clomiphene citrate regimen (Active Comparator)
  Interventions: Drug: Clomiphene citrate regimen

INTERVENTIONS:
Drug: Extended letrozole regimen — Letrozole (Femara; Novartis pharma AG, Basle, Switzerland) 2.5mg /day is administered from cycle day 1 to 9 .
  Human chorionic gonadotropin (Pregnyl; N.V. Organon, Oss, Holland) ( 10.000 IU/I.M ) is administered to trigger ovulation when at least one follicle measures more than 18mm in mean diameter .Intrauterine insemination is performed 36 - 40 hours after HCG injection .
  Starting from cycle day 9 , ultrasound scans are repeated daily to monitor follicle growth . Serum estradiol and endometrial thickness are measured on the day of HCG administration.
  Serum B-subunit HCG is measured 2 weeks after IUI to diagnose pregnancy .
  Other Names: letrozole 2.5mg/day from cycle day 1 to 9
  Arms: Extended letrozole regimen
Drug: Clomiphene citrate regimen — Clomiphene citrate(Clomid; Aventis pharma S.AE, Global Napi pharmaceuticals, Cairo, Egypt) 100 mg/day is administered from cycle day 3 to 7.
  Human chorionic gonadotropin (Pregnyl; N.V. Organon, Oss, Holland) ( 10.000 IU/I.M ) is administered to trigger ovulation when at least one follicle measures more than 18mm in mean diameter .Intrauterine insemination is performed 36 - 40 hours after HCG injection .
  Starting from cycle day 9 , ultrasound scans are repeated daily to monitor follicle growth . Serum estradiol and endometrial thickness are measured on the day of HCG administration.
  Serum B-subunit HCG is measured 2 weeks after IUI to diagnose pregnancy .
  Other Names: Clomiphene citrate 100mg/day from cycle day 3 to 7
  Arms: Clomiphene citrate regimen

SUMMARY:
The aim of this randomized controlled trial is to compare the efficacy of extended letrozole regimen (2.5mg/day from cycle day 1 to 9) with clomiphene citrate (100 mg/day from cycle day 3 to 7) in women with unexplained infertility undergoing superovulation and intrauterine insemination .

DETAILED DESCRIPTION:
Unexplained infertility is one of the most frequent infertility diagnoses encountered by the gynaecologists . Several studies reported that 10 to 20% of infertile couples have unexplained infertility .

Superovulation and intrauterine insemination (IUI) is an effective treatment for couples with unexplained infertility . Superovulation increases the probability of pregnancy by increasing the number of oocytes suitable for fertilization or by correcting any subtle defect in ovulation . Furthermore, IUI increases the concentration of active motile sperms reaching the fallopian tube and overcomes male factors or cervical factors of infertility not detected by conventional tests .

For more than four decades , clomiphene citrate has been the first line therapy used for induction of ovulation in women with anovulatory infertility and for superovulation in couples with unexplained infertility, mild endometriosis and mild male factor of infertility . Clomiphene citrate is cheap , orally administered , requires no frequent monitoring and associated with very low risk of high-order multiple gestation and severe ovarian hyperstimulation syndrome . However , clomiphene citrate causes long lasting depletion of estrogen receptors and therefore exerts antiestrogenic effect on estrogen target tissues as endocervical mucosa and endometrium .Several studies revealed the clomiphene citrate has a deleterious effect on cervical mucous quantity and quality and endometrial development resulting in endometrial thinning , luteal phase defect ,decreased uterine flow and implantation failure .

During the past decade, letrozole (aromatase inhibitor approved by FDA for the treatment of postmenopausal women with breast cancer ) has been successfully used in induction of ovulation in anovulatory patients with polycystic ovary syndrome and in augmentation of ovulation in ovulatory women . In contrast to clomiphene citrate , letrozole is rapidly eliminated from the body and does not deplete estrogen receptors and therefore has no antiestrogenic effects on endometrium or endocervical mucosa .

Several studies revealed that letrozole can be used as an alternative to clomiphene citrate for superovulation in patients with unexplained infertility . A metaanalysis of seven randomized controlled trials comparing aromatase inhibitors ( letrozole or anastrozole ) with clomiphene citrate in patients with unexplained infertility revealed that the pregnancy rate was comparable between both management options .

The optimal dose and duration of letrozole administration for superovulation in patients with unexplained infertility is still not clear. In various studies reporting the use of letrozole for the superovulation , letrozole was administrated from cycle 3 to 7 with daily dose ranging from 2.5 to 7.5 mg .In a randomized controlled trial , AI-Fadhli et al reported that the pregnancy rate was significantly higher in patients with unexplained infertility treated with 5 mg compared to those treated with 2.5 mg . On the other hand, a randomized controlled trial comparing three doses of letrozole (2.5,5,7.5 mg/day)in the management of patients with unexplained infertility revealed that the pregnancy rates were comparable between the three groups .

The aim of this randomized controlled trial is to compare the efficacy of extended letrozole regimen (2.5mg/day from cycle day 1 to 9) with clomiphene citrate (100 mg/day from cycle day 3 to 7) in women with unexplained infertility undergoing superovulation and intrauterine insemination .

ELIGIBILITY:
Inclusion Criteria:

* Patients with unexplained infertility
* Age between 18 - 37 years
* Period of infertility > 1 year
* Patent Fallopian tubes detected by hysterosalpingography and/or laparoscopy
* Normal basal luteinizing hormone (LH), follicle stimulating hormone (FSH) and prolactin concentrations
* Normal recent semen analysis (according to World Health Organization criteria)

Exclusion Criteria:

* FSH> 10 IU/L
* Irregular menstrual cycles
* Polycystic ovary syndrome
* Endometriosis
* Endocrinologic disorders
* Systemic disease contraindicating pregnancy
* Previous IUI cycles
* liver or kidney diseases

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 214 (Actual)
Dates: Start 2008-09; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 5 weeks after intrauterine insemination
  Presence of intrauterine gestational sac detected by transvaginal ultrasound

SECONDARY OUTCOMES:
Ongoing Pregnancy Rate | 18 weeks after intrauterine insemination
  Pregnancies continued beyond 20 weeks gestation

CONTACTS AND LOCATIONS:
Overall Officials: Usama M Fouda, M.D, PhD, Study Chair — Cairo University; Ahmed M Sayed, M.D, PhD, Study Director — Cairo University
Locations (2):
- Egypt (2):
  - Ahmed Elgazzar hospital, Cairo
  - Cairo university hospital, Cairo

REFERENCES:
- [Background] Badawy A, Mosbah A, Tharwat A, Eid M. Extended letrozole therapy for ovulation induction in clomiphene-resistant women with polycystic ovary syndrome: a novel protocol. Fertil Steril. 2009 Jul;92(1):236-9. doi: 10.1016/j.fertnstert.2008.04.065. Epub 2008 Aug 15. PMID 18706549
- [Background] Badawy A, Elnashar A, Totongy M. RETRACTED: Clomiphene citrate or aromatase inhibitors for superovulation in women with unexplained infertility undergoing intrauterine insemination: a prospective randomized trial. Fertil Steril. 2009 Oct;92(4):1355-1359. doi: 10.1016/j.fertnstert.2008.06.013. Epub 2008 Aug 9. PMID 18692823
- [Derived] Fouda UM, Sayed AM. Extended letrozole regimen versus clomiphene citrate for superovulation in patients with unexplained infertility undergoing intrauterine insemination: a randomized controlled trial. Reprod Biol Endocrinol. 2011 Jun 21;9:84. doi: 10.1186/1477-7827-9-84. PMID 21693030